CLINICAL TRIAL: NCT00002986
Title: Phase I Treatment of Adults With Primary Malignant Glioma With Topotecan (NSC #609699) Plus BCNU (NSC #409962)
Brief Title: Chemotherapy in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0224; DUMC-000224-01-1R4; DUMC-000224-00-2R3; DUMC-0348-99-2R2; DUMC-223-97-2; DUMC-229-98-2R1; SB-DUMC-229-98-2R1; NCI-G97-1242; CDR0000065521 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Carmustine; Topotecan

INTERVENTIONS:
Drug: carmustine
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of topotecan plus carmustine in patients with recurrent primary malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of topotecan administered in combination with a fixed dose of carmustine.
* Determine the toxic effects of topotecan and carmustine in patients with recurrent primary malignant glioma.

OUTLINE: Topotecan is administered by an ambulatory infusion pump for 72 hours each week. Topotecan dose escalation is carried out in cohorts of three patients. Dose escalation is continued until toxic effects or disease progression is observed in these patients. Carmustine is administered over 1 hour every 6 weeks, on the same day as the first topotecan dose for that week.

Three patients will be treated at an initial dose level of topotecan, and if one of these patients experience dose limiting toxicity (DLT), an additional

3 patients must be treated at this dose level without further DLT in order for dose escalation to proceed. The MTD is the highest dose at which DLT occurs in no more than 1 of 6 patients.

Patients are evaluated after every 6 week cycle.

PROJECTED ACCRUAL: An estimated 18-36 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent primary malignant glioma

  * Measurable recurrent or residual primary central nervous system neoplasm confirmed by MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance Status:

* Karnofsky at least 60%

Hematopoietic:

* Hematocrit greater than 29%
* ANC greater than 1,500/mm^3
* Platelet count greater than 125,000/mm^3

Hepatic:

* SGOT less than 1.5 times upper limit of normal (ULN)
* Bilirubin less than 1.5 times ULN

Renal:

* Creatinine less than 1.5 mg/dL
* BUN less than 25 mg/dL

Other:

* Not pregnant
* Effective contraceptive method must be used for the duration of the study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy within 6 weeks of study
* No prior topotecan or carmustine treatment failure
* No more than 1 prior chemotherapy regimen

Endocrine therapy:

* Patients taking corticosteroids must be on stable dose for at least 2 weeks prior to study and the dose should not escalate over entry level

Radiotherapy:

* No prior radiotherapy within 6 weeks of study

Surgery:

* No prior surgical resection within 3 weeks of study

Other:

* No concurrent medication that may interfere with study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1997-02; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (2):
- United States (2):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee